CLINICAL TRIAL: NCT00617994
Title: An Open Label, Safety, Tolerability, Pharmacokinetic (PK), Pharmacodynamic (PD) and Preliminary Efficacy Study of Ruxolitinib When Applied to Patients With Plaque Psoriasis Involving 2 - 20% Body Surface Area (BSA).
Brief Title: Open Label, Safety and Efficacy Study of Topical Investigational Drug to Treat Patients With Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-202
Record Dates: First submitted 2008-01-21; First posted 2008-02-18 (Estimated); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Patients with active stable plaque psoriasis treated with topical cream application on lesions involving a small percent BSA.
  Interventions: Drug: Ruxolitinib
- Group B (Experimental): Patients with active stable plaque psoriasis treated with topical cream application on lesions involving a larger percent BSA than Cohort 1.
  Interventions: Drug: Ruxolitinib
- Group C (Experimental): Patients with active stable plaque psoriasis treated with topical cream application on lesions involving a larger percent BSA than Cohort 2.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib 1.5% cream BID for 28 days
  Other Names: INCB018424

SUMMARY:
This will be an open label study of ruxolitinib topical cream applied to 2 - 20% BSA in patients with active, stable plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have psoriatic lesions measuring protocol specific BSA

Exclusion Criteria:

* Lesions solely involving the palms of the hands, the soles of the feet, the intertriginious areas, the scalp or the face
* Pustular psoriasis or erythroderma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-08-31 (Actual); Primary Completion 2009-04-30 (Actual); Study Completion 2009-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Williams, MD, Study Director — Incyte Corporation
Locations (4):
- United States (4):
  - Fridley, Minnesota
  - Rochester, New York
  - Austin, Texas
  - College Station, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 study centers in the United States from 08 November 2007 to 13 April 2009. This study is completed.
Pre-assignment Details: A total of 25 participants with active but stable plaque psoriasis were enrolled in the dose-escalation study.
Groups:
- Cohort A: 2% to 7% of BSA treated BID with INCB018424 1.5% cream
- Cohort B: 8% to 13% of BSA treated BID with INCB018424 1.5% cream
- Cohort C: 14% to 20% of BSA treated QD with INCB018424 1.5% cream
- Cohort D: 14% to 20% of BSA treated BID with INCB018424 1.0% cream
- Cohort E: 14% to 20% of BSA treated BID with INCB018424 1.5% cream
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Cohort E
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT: The intent-to-treat (ITT) population included all enrolled participants who applied INCB018424 cream at least once and had a predose and at least one post-dose lesion assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Cohort E | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (6.22) | 32.4 (7.57) | 43.2 (13.94) | 46.2 (12.21) | 42.8 (18.16) | 40.5 (12.36)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 5 | 3 | 4 | 4 | 4 | 20
  Female | 0 | 2 | 1 | 1 | 1 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian/Alaskan Native White | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian/Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  White or Caucasian | 4 | 5 | 5 | 5 | 3 | 22
  Other | 1 | 0 | 0 | 0 | 2 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 1 | 4
  Not Hispanic or Latino | 4 | 4 | 4 | 5 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment of Emergent Adverse Events
Description: Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment
Time Frame: Approximately 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Participants | 2 | 4 | 2 | 1 | 2

2. Primary Outcome: Pharmacokinetics Parameter : Skin Flux of INCB018424
Description: The INCB018424 skin flux was estimated from the overall mean steady-state plasma concentrations for each subject in this study and the estimated systemic clearance of INCB018424 following oral-dose administration in another study.
Time Frame: Days 1, 4, 8, 15, 22, and 28-30
Measure: Mean (Standard Deviation); unit: ng/cm^2/h
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
ng/cm^2/h | 180 (126) | 131 (92) | 60 (43) | 151 (126) | 152 (74)

3. Primary Outcome: Pharmacokinetics Parameter: Bioavailability of INCB018424
Description: The INCB018424 bioavailability was estimated from the overall mean steady-state plasma concentrations for each subject in this study and the estimated systemic clearance of INCB018424 following oral-dose administration in another study.
Time Frame: Approximately one month: Days 1, 4, 8, 15, 22, and 28
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
percentage | 3.8 (2.5) | 4.1 (3.4) | 3.4 (1.9) | 3.9 (1.3) | 5.2 (1.9)

4. Secondary Outcome: Psioriatic Lesion Severity: Change in Total Lesion Score for the Target Lesion Compared to Baseline
Description: Changes in total lesion scores were compared to baseline score. Lesions were compared between active treated areas INCB018424 and control areas of the same subject (within-subject comparisons) using one sample t-test. Total lesion score was calculated as the sum of the scores for Thickness (T), erythema (E), and scaling (S) for the target and control lesions. All individual scores use a 5-point scale ranging from 0 (none) to 4 (severe) with increasing score reflecting increased lesion severity. These ratings are then added to create a total score ranging from 0 to 12.
Time Frame: Approximately 2 months (Days 1, 8, 15, 22, 28 and up to an additional 28 day Follow-Up)
Measure: Mean (95% Confidence Interval); unit: Change in Total Score
Groups:
- Cohort A: Control Lesion; Cohort B: Control Lesion; Cohort C: Control Lesion; Cohort D: Control Lesion; Cohort E: Control Lesion: Control Lesions were not treated.
Arm/Group | Cohort A: Control Lesion | Cohort A | Cohort B: Control Lesion | Cohort B | Cohort C: Control Lesion | Cohort C | Cohort D: Control Lesion | Cohort D | Cohort E: Control Lesion | Cohort E
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Change in Total Score
  Day 8 | .4 [0 to 2] | -1.4 [-4 to 1] | -0.8 [-3 to 0] | -4.0 [-6 to -2] | -0.2 [-1 to 0] | -1.2 [-5 to 1] | -0.2 [-2 to 1] | -1.2 [-2 to 0] | 0.2 [0 to 1] | -2.8 [-5 to 2]
  Day 15 | 0.2 [-1 to 2] | -3.2 [-5 to -2] | -2.00 [-4 to -1] | -4.2 [-7 to -2] | -0.6 [-2 to 0] | -2.6 [-7 to 0] | 0.8 [0 to 2] | -0.8 [-4 to 0] | -0.8 [-4 to 0] | -3.6 [-6 to -2]
  Day 22 | 1.0 [0 to 2] | -2.8 [-6 to 0] | -1.8 [-4 to -1] | -5.0 [-7 to -2] | -2.8 [-6 to 0] | -3.6 [-7 to -1] | 1.0 [0 to 3] | -2.8 [-6 to -1] | -0.4 [-3 to 1] | -3.6 [-7 to -2]
  Day 28 | 0.8 [-1 to 2] | -3.4 [-6 to -2] | -2.0 [-4 to 0] | -5.4 [-7 to -3] | -3.6 [-8 to 0] | -4.4 [-8 to -2] | 0.6 [0 to 1] | -3.6 [-5 to -2] | -1.2 [-6 to 0] | -3.8 [-7 to -2]
  Follow-up | 1.2 [0 to 2] | -1.2 [-4 to 1] | 1.0 [-3 to 1] | -3.6 [-6 to 0] | -4.2 [-9 to 0] | -3.2 [-9 to 1] | 0.6 [-1 to 2] | -1.0 [-3 to 0] | -2.0 [-6 to 0] | -2.8 [-7 to 0]

5. Secondary Outcome: Mean Change in Psoriatic Lesion Area
Description: The target and control lesion areas were determined in an objective manner on Day 1 and Day 28 based on a tracing of the perimeter of the lesions on transparency film and measurement of the area.
Time Frame: Days 1 and 28
Measure: Mean (Standard Deviation); unit: cm^2
Groups:
- Cohort D: Control Lesion; Control E: Control Lesion: Control lesions were untreated.
Arm/Group | Cohort A: Control Lesion | Cohort A | Cohort B: Control Lesion | Cohort B | Cohort C: Control Lesion | Cohort C | Cohort D: Control Lesion | Cohort D | Control E: Control Lesion | Cohort E
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5
cm^2 | -2.20 (23.993) | -237.76 (240.500) | -15.94 (38.247) | -620.56 (714.829) | 0.40 (11.336) | -1267.78 (1009.159) | -9.02 (10.346) | -871.12 (1062.346) | -12.32 (23.283) | -823.78 (313.733)

6. Secondary Outcome: Mean Change in Physicians Global Assessment Score
Description: The PGA was an overall assessment of each participant's plaque psoriasis. The assessment was recorded using a scale that ranged from 0 (clear) to 6 (most severe) in whole-unit increments.
  Note that, for analysis purposes, the scale was adjusted to range from 1 (clear) to 7 (most severe) to allow for the evaluation of mean scores.
Time Frame: Approximately 2 months: Days 1, 8, 15, 22, 28 and follow-up approximately one month later
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Score
  Screening | 4.4 (0.55) | 4.4 (0.89) | 4.2 (0.45) | 4.4 (0.55) | 4.0 (0.00)
  Day 1 | 4.0 (0.00) | 4.4 (0.89) | 4.2 (0.45) | 4.4 (0.55) | 4.0 (0.00)
  Day 8 | 3.4 (0.55) | 3.6 (0.55) | 4.0 (0.71) | 4.2 (0.45) | 3.0 (0.00)
  Day 15 | 2.6 (0.55) | 3.2 (0.84) | 3.8 (0.84) | 3.8 (0.45) | 2.6 (0.55)
  Day 22 | 2.4 (0.55) | 3.0 (0.71) | 3.6 (0.89) | 3.2 (0.45) | 2.6 (0.55)
  Day 28 | 2.4 (0.55) | 2.6 (0.89) | 3.4 (0.55) | 3.0 (0.71) | 2.4 (0.55)
  Follow-up | 3.4 (0.89) | 3.4 (0.89) | 3.2 (1.30) | 4.0 (0.71) | 3.2 (0.45)

7. Primary Outcome: Pharmacokinetics Parameter: Plasma Concentrated Steady State (CSS) of INCB018424
Description: All observed INCB018424 plasma concentrations from Days 8, 15, 22, and 28 were averaged to obtain an overall mean exposure for each subject. Samples were taken pre-dose and approximately one hour post-dose.
Time Frame: Approximately one month: Days 1, 4, 8, 15, 22, and 28
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
nM | 7.00 (2.10) | 28.38 (13.10) | 24.41 (10.07) | 34.97 (20.44) | 60.98 (73.85)

ADVERSE EVENTS:
Groups:
- Cohort A: 2 to 7% of BSA treated BID with INCB018424 1.5% cream
- Cohort B: 8 to 13% of BSA treated BID with INCB018424 1.5% cream BID
- Cohort C: 14 to 20% of BSA treated QD with INCB018424 1.5% cream QD
- Cohort D: 14-20% of BSA with INCB018424 1.0% cream BID
- Cohort E: 14 to 20% of BSA treated BID with INCB018424 1.5% cream BID
- Total: Total
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Cohort E | Total
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 1/5 | 0/5 | 0/5 | 1/25
Other Adverse Events (participants affected / at risk) | 2/5 | 4/5 | 2/5 | 1/5 | 2/5 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=5) | Cohort B (N=5) | Cohort C (N=5) | Cohort D (N=5) | Cohort E (N=5) | Total (N=25)
Schizophrenia, paranoid type (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=5) | Cohort B (N=5) | Cohort C (N=5) | Cohort D (N=5) | Cohort E (N=5) | Total (N=25)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reticulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement